CLINICAL TRIAL: NCT00608049
Title: Optimal Macronutrient Intake - Carbohydrate
Brief Title: Effect of Amount and Type of Dietary Carbohydrates on Risk for Cardiovascular Heart Disease and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank M. Sacks, Frank M. Sacks, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 481; R01HL084568 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Overweight; Cardiovascular Diseases
Keywords: Blood Pressure; Diabetes; Nutrition; Dietary Carbohydrate; Lipoproteins; Insulin Resistance
MeSH Terms: conditions — Overweight; Cardiovascular Diseases; Diabetes Mellitus; Insulin Resistance | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: high carbohydrate/high GI, high carbohydrate/low GI, low carbohydrate/high GI, and low carbohydrate/low GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 2 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: high carbohydrate/high GI, high carbohydrate/low GI, low carbohydrate/low GI, and low carbohydrate/high GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 3 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: high carbohydrate/low GI, high carbohydrate/high GI, low carbohydrate/high GI, and low carbohydrate/low GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 4 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: high carbohydrate/low GI, high carbohydrate/high GI, low carbohydrate/low GI, and low carbohydrate/high GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 5 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: low carbohydrate/high GI, low carbohydrate/low GI, high carbohydrate/high GI, and high carbohydrate/low GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 6 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: low carbohydrate/high GI, low carbohydrate/low GI, high carbohydrate/low GI, and high carbohydrate/high GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 7 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: low carbohydrate/low GI, low carbohydrate/high GI, high carbohydrate/high GI, and high carbohydrate/low GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet
- 8 (Experimental): Participants will follow four diet plans, each for a period of 5 weeks, in the following order: low carbohydrate/low GI, low carbohydrate/high GI, high carbohydrate/low GI, and high carbohydrate/high GI
  Interventions: Behavioral: High carbohydrate and low glycemic index (GI) diet; Behavioral: Low carbohydrate and low GI diet; Behavioral: High carbohydrate and high GI diet; Behavioral: Low carbohydrate and high GI diet

INTERVENTIONS:
Behavioral: High carbohydrate and low glycemic index (GI) diet — The high carbohydrate and low GI diet will require 58% of daily calories to be from carbohydrates and will be composed of meals with a GI of less than 45 on the glucose scale.
Behavioral: Low carbohydrate and low GI diet — The low carbohydrate and low GI diet will require 40% of daily calories to be from carbohydrates and will be composed of meals with a GI of less than 45 on the glucose scale.
Behavioral: High carbohydrate and high GI diet — The high carbohydrate and high GI diet will require 58% of daily calories to be from carbohydrates and will be composed of meals with a GI of greater than 65 on the glucose scale.
Behavioral: Low carbohydrate and high GI diet — The low carbohydrate and high GI diet will require 40% of daily calories to be from carbohydrates and will be composed of meals with a GI of greater than 65 on the glucose scale.

SUMMARY:
Cardiovascular disease (CVD) and diabetes are health conditions that are strongly influenced by a person's diet. Although the best diet to prevent CVD and diabetes is uncertain, reducing intake of saturated and transunsaturated fats is known to help lower cardiovascular risk. However, even diets low in these fats can vary widely in other energy providing nutrients, particularly carbohydrates. This study will determine the effects of a higher versus lower carbohydrate diet, each with a high or low glycemic index (GI) composition, on risk factors for CVD and diabetes.

DETAILED DESCRIPTION:
A healthy diet can have a remarkable effect on a person's overall health. Research has consistently confirmed the association between diet and serious health problems, including heart disease, diabetes, high blood pressure, and gastrointestinal disorders. Most healthy diets aimed at disease prevention promote a low intake of fats, but the optimal diet to prevent CVD and related disorders is uncertain. Recent emphasis has turned to the influence of carbohydrate consumption on risk of CVD and diabetes. Carbohydrates comprise a wide range of foods, which are categorized by their absorption rate, also known as glycemic index (GI). There is much current debate over how the level and type of dietary carbohydrates affect cardiovascular health. This study will determine the effects of a higher versus lower carbohydrate diet, each with a high or low GI composition, on risk factors for CVD and diabetes.

Potential participants will attend three screening visits that will include questionnaires, clinical measurements, and blood and urine tests. Participants will then undergo an 8-day run-in phase to become familiar with the feeding patterns of four different diets: high carbohydrate with high GI, high carbohydrate with low GI, low carbohydrate with high GI, or low carbohydrate with low GI. During the run-in, participants will be provided all of their food, snacks, and calorie-containing beverages. Participants will also complete a daily food diary, symptoms questionnaire, medical and social history, and daily weigh-in. After meeting with a dietician to review progress, eligible participants will be randomly assigned to one of eight sequences of the four diet plans.

Participants will follow each of the four diet plans for 5 weeks, with a period of at least 2 weeks separating each plan. During each dieting period, participants will be provided all of their food and snacks and most beverages. All participants will be required to eat at least one on-site meal per day, 5 days per week. Participants will keep a daily food diary and will undergo weekly blood pressure measurements for the first 3 weeks of each dieting period. Assessments will occur in the fifth week of each of the four dieting periods and will include symptoms and satiety questionnaires, blood pressure measurements, and a blood draw. One month following the completion of the last dieting period, participants will receive nutritional counseling on the prevention of CVD.

ELIGIBILITY:
Inclusion Criteria:

* SBP of 120 to 159 mmHg and DBP less than 100 mmHg at study entry (mean over three screening visits) (note: participants with stage 2 hypertension [SBP greater than 160 mmHg or DBP greater than 100 mmHg] based on the mean over three screening visits will be excluded, as will participants with a mean SBP greater than 170 mmHg or DBP greater than 105 mmHg at any one visit)
* Overweight or obese, as defined by a body mass index (BMI) greater than 25 kg/m2
* Willing to eat at least one on-site meal per day, 5 days per week, and willing to eat study diets and nothing else during controlled feeding periods

Medication Exclusion Criteria:

* Symptomatic ischemic heart disease (e.g., angina pectoris)
* Regular use of medications that raise or lower BP during the 2 months prior to study entry
* Use of a lipid lowering agent in the 3 weeks prior to study entry
* Unstable dose of hormone replacement therapy, thyroid hormone replacement therapy, and psychotropic medications known to cause weight gain or affect the outcome variables (unstable is defined as a change in dose within 2 months of study entry)
* Use of insulin, oral hypoglycemic agent, lithium, oral corticosteroid, anti-psychotic drugs, weight loss medications, nitrate, or digitalis

Medical History Exclusion Criteria:

* Active or prior CVD (e.g., stroke, heart attack, percutaneous transluminal coronary angioplasty, coronary artery bypass graft, congestive heart failure, symptomatic ischemic heart disease [angina], or arteriosclerotic cardiovascular disease-related therapeutic procedure)
* Diabetes mellitus
* Cancer diagnosis or treatment in the 2 years prior to study entry (note: people with non-melanoma skin cancer, localized breast cancer, or localized prostate cancer can enroll if they did not require systemic chemotherapy)
* Active inflammatory bowel disease, malabsorption, or major gastrointestinal resection
* Renal insufficiency as determined by a serum creatinine greater than 1.2 mg/dL for women or greater than 1.4 mg/dL for men (these participants can enroll if their estimated glomerular filtration rate is greater than 40 mL/min by either the Cockcroft-Gault equation or the simplified Modification of Diet in Renal Disease equation)
* Emergency room visit or hospital stay for asthma or chronic obstructive pulmonary disease in the 6 months prior to study entry
* Any serious illness not otherwise specified that would interfere with participation

Laboratory Exclusion Criteria:

* Fasting LDL cholesterol greater than 220 mg/dL and triglycerides greater than 750 mg/dL
* Fasting blood glucose greater than 125 mg/dL
* Serum transaminase greater than 2 times the upper range of normal, or a clinical diagnosis of hepatitis

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP), Low Density Lipoproteins (LDL) cholesterol, High Density Lipoproteins (HDL) cholesterol, triglycerides, and insulin sensitivity | Measured at Week 5 of each dieting period

SECONDARY OUTCOMES:
Diastolic blood pressure (DBP); apolipoproteins B, CIII, A-I, and Very Low Density Lipoproteins (VLDL); and LDL with apolipoprotein CIII | Measured at Week 5 of each dieting period
Beta cell response, glucose effectiveness, and fructosamine; postprandial glucose, insulin, lipids, and hormone levels | Measured at Week 5 of each dieting period
Overall CVD risk using risk equations | Measured at Week 5 of each dieting period

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Sacks, MD, Principal Investigator — Harvard University; Lawrence J. Appel, MD, Study Director — Johns Hopkins Medical Institutions, Baltimore
Locations (2):
- United States (2):
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Harvard T. H. Chan School of Public Health, Boston, Massachusetts

REFERENCES:
- [Derived] Wu Y, Juraschek SP, Hu JR, Mueller NT, Appel LJ, Anderson CAM, Miller ER. Higher Carbohydrate Amount and Lower Glycemic Index Increase Hunger, Diet Satisfaction, and Heartburn in Overweight and Obese Adults in the OmniCarb Randomized Clinical Trial. J Nutr. 2021 Aug 7;151(8):2477-2485. doi: 10.1093/jn/nxab128. PMID 34049396
- [Derived] Hu JR, Wu Y, Sacks FM, Appel LJ, Miller Iii ER, Young JH, Juraschek SP. Effects of carbohydrate quality and amount on plasma lactate: results from the OmniCarb trial. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001457. doi: 10.1136/bmjdrc-2020-001457. PMID 32868311
- [Derived] Juraschek SP, Miller ER 3rd, Selvin E, Carey VJ, Appel LJ, Christenson RH, Sacks FM. Effect of type and amount of dietary carbohydrate on biomarkers of glucose homeostasis and C reactive protein in overweight or obese adults: results from the OmniCarb trial. BMJ Open Diabetes Res Care. 2016 Nov 14;4(1):e000276. doi: 10.1136/bmjdrc-2016-000276. eCollection 2016. PMID 27933186
- [Derived] Juraschek SP, Chang AR, Appel LJ, Anderson CA, Crews DC, Thomas L, Charleston J, Miller ER 3rd. Effect of glycemic index and carbohydrate intake on kidney function in healthy adults. BMC Nephrol. 2016 Jul 8;17(1):70. doi: 10.1186/s12882-016-0288-5. PMID 27391484
- [Derived] Juraschek SP, McAdams-Demarco M, Gelber AC, Sacks FM, Appel LJ, White KJ, Miller ER 3rd. Effects of Lowering Glycemic Index of Dietary Carbohydrate on Plasma Uric Acid Levels: The OmniCarb Randomized Clinical Trial. Arthritis Rheumatol. 2016 May;68(5):1281-9. doi: 10.1002/art.39527. PMID 26636424
- [Derived] Sacks FM, Carey VJ, Anderson CA, Miller ER 3rd, Copeland T, Charleston J, Harshfield BJ, Laranjo N, McCarron P, Swain J, White K, Yee K, Appel LJ. Effects of high vs low glycemic index of dietary carbohydrate on cardiovascular disease risk factors and insulin sensitivity: the OmniCarb randomized clinical trial. JAMA. 2014 Dec 17;312(23):2531-41. doi: 10.1001/jama.2014.16658. PMID 25514303